CLINICAL TRIAL: NCT00165906
Title: A Pilot Study Examining Thrombin Generation in the Neonatal Population
Brief Title: Thrombin Generation in Neonates
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Nina Guzzetta, M.D., Assistant Professor of Anesthesiology, Emory University
Other Study IDs: IRB00000300
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Blood Coagulation Disorders
Keywords: neonates; cardiac; non-cardiac; surgery; anticoagulation
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample is obtained to measure the thrombin level.
Oversight: Data Monitoring Committee: No

SUMMARY:
Children having open heart surgery must be on a heart-lung bypass machine. It is essential that the blood in the heart-lung machine does not clot. This is accomplished by giving a drug called heparin, a "blood thinner".

The process of making a clot involves a lot of steps. One of the steps involves a protein called thrombin. Heparin acts on thrombin to keep blood from clotting. A technique has been developed to measure the blood's ability to generate thrombin. The bloods's ability to generate thrombin is measured by a thrombin generation curve (TGC). This curve would be very helpful to know when choosing the dose of heparin. We haven't found any studies using TGC in babies less than a month old.

We want to do a study comparing the TGC in 10 newborns without a heart defect to the TGC in 10 newborns with a congenital heart defect. To do this we will need one sample of blood. the sample we need is 3 cc which is a little more than 1/2 teaspoon. The blood sample for both groups is to be taken from the intravenous catheter (IV) the child will have placed for surgery. The newborns without a heart defect will be children having surgery for a non-cardiac problem.

DETAILED DESCRIPTION:
Neonates are unique due to maturational differences in their coagulation systems. During the first few months of life, distinct differences exist between the coagulation system of a neonate and that of an adult including differences between the concentration of coagulation proteins, the ability to generate thrombin and the ability to inhibit thrombin once it is formed (1). One important coagulant protein that is quantitatively deficient in the first several months of life is prothrombin. In the coagulation cascade, prothrombin is converted into thrombin, a major regulator of hemostasis. In healthy newborns mean prothrombin values are less than 70% of adult mean values (1), and investigators have found that neonatal prothrombin level is directly proportional to the amount of thrombin generated (1). In fact, the impaired ability of newborn plasma to generate thrombin in the face of deficient prothrombin has been shown to be similar to adults who are being treated therapeutically with an anticoagulant (2). Therefore, low prothrombin levels in neonates have important implications when considering anticoagulant therapy.

For neonates with congenital heart disease presenting for cardiac surgery, anticoagulation for cardiopulmonary bypass (CPB) is necessary to prevent clotting as blood comes into contact with the unphysiologic surfaces of the extracorporeal circuit. This is achieved by the use of high dose heparin, which is used to inhibit the formation and activation of thrombin. Since neonatal prothrombin levels are low, rendering them unable to generate large amounts of thrombin, neonates with congenital heart disease requiring anticoagulation for CPB have historically been considered heparin sensitive (3). However, in a recent investigation conducted by this group, elevated baseline levels of thrombin production and activity were consistently found in neonates presenting for cardiac surgery (4). Additionally, despite routine heparin dosing, elevated markers of thrombin production were also found in these neonates during CPB when compared to their adult counterparts (4). Perhaps the assumption that neonates with congenital heart disease are similar to other healthy neonates in their impaired ability to generate thrombin is incorrect. Contact activation may occur preoperatively from the presence of indwelling umbilical catheters and central lines or from interventional manipulations in the cardiac catheterization lab and stimulate their coagulation systems to generate more thrombin than anticipated. Elevated thrombin levels in neonates presenting for cardiac surgery would consequently have important implications in determining the optimal heparin dose needed to provide adequate anticoagulation for CPB.

A technique has been developed to monitor the thrombin generating capacity of plasma (5). A thrombin generation curve (TGC) can be constructed from a sample of plasma and the area under the TGC, called the endogenous thrombin potential (ETP), is a good indicator of the coagulability of the sample. Currently, we have found no published data addressing the TGC in the neonatal population. Therefore, we propose a prospective study between neonates with congenital heart disease presenting for cardiac surgery and other healthy neonates to compare their respective abilities to generate thrombin by measuring TGCs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective cardiac surgery scheduled at Children's Healthcare of Atlanta as a first time procedure OR patients undergoing elective non-cardiac surgery scheduled at Children's Healthcare of Atlanta (control group)
2. Patients within the appropriate age group, i.e. less than 1 month old
3. Parents or legal guardian willing for the child to participate and able to sign the provided informed consent -

Exclusion Criteria:

1. Patients undergoing any emergent procedure/surgery
2. Patients who are being administered preoperative anticoagulant therapy
3. Patients with a known coagulation defect or coagulopathy
4. Patients who are premature, i.e. less than 37 weeks gestational age
5. Patient who are greater than 1 month of age
6. Parents or legal guardian are unwilling or unable to sign the provided informed consent
7. Patients who in the opinion of the investigators should not be included in the study

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study patients will be obtained from Children's Healthcare of Atlanta at Egleston. The study patients will be in the pre-operative clinic, Cardiac Intensive Care Unit or the Cardiac Stepdown Unit.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina A Guzzetta, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kern FH, Morana NJ, Sears JJ, Hickey PR. Coagulation defects in neonates during cardiopulmonary bypass. Ann Thorac Surg. 1992 Sep;54(3):541-6. doi: 10.1016/0003-4975(92)90451-9. PMID 1510523
- [Background] Guzzetta NA, Miller BE, Todd K, Szlam F, Moore RH, Tosone SR. An evaluation of the effects of a standard heparin dose on thrombin inhibition during cardiopulmonary bypass in neonates. Anesth Analg. 2005 May;100(5):1276-1282. doi: 10.1213/01.ANE.0000149590.59294.3A. PMID 15845669